CLINICAL TRIAL: NCT01668082
Title: An Investigation of Brain Tumor Metabolism in Patients Undergoing Surgical Resection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Elizabeth Maher, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU 062010-157
Record Dates: First submitted 2012-06-12; First posted 2012-08-17 (Estimated); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Brain Mass
Keywords: Patients with newly identified brain mass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- surgical resection of a brain tumor (Experimental): The patient will undergo surgical removal of the tumor after infusion of 13C-glucose using standard neurosurgical technique, including frameless stereotaxy for surgical navigation, and microsurgical technique.
  --------------------------------------------------------------------------------
  Interventions: Procedure: surgical resection of a brain tumor

INTERVENTIONS:
Procedure: surgical resection of a brain tumor — The patient will undergo surgical removal of the tumor after infusion of 13C-glucose using standard neurosurgical technique, including frameless stereotaxy for surgical navigation, and microsurgical technique.

SUMMARY:
The study is designed to use infusion of a non-radioactive, naturally occurring isotope of glucose (13C) in patients undergoing surgical resection for a newly identified brain mass to obtain the metabolic phenotype of the tumor, and correlate it with the histopathological diagnosis. In each patient, 13C NMR spectral analysis of tumor extracts will be obtained after intraoperative infusion of [U-13C]glucose or [1,2-13C]glucose. Whenever feasible, patients will undergo 3 preoperative imaging studies - 18FDG-PET, diffusion tensor imaging with 1H-spectroscopy on 3T MR scanner, and ultra high resolution MR imaging on the 7T MR scanner. The results of these imaging studies will be correlated with the metabolic phenotype to generate a comprehensive non-invasive view of the tumor with the goal of identifying infiltrative, metabolically active tumor cells within the brain. In addition, a comprehensive molecular profile of the tumor will be obtained and enable a genotype-metabolic phenotype comparative analysis.

Correlative Translational Research The investigators will obtain tumor tissue from each patient for comprehensive molecular analysis (array CGH, expression profiling, methylation profiling) which will be correlated with tumor histology, the metabolites identified by 1H-MR spectroscopy and the 13Cglucose metabolic profile. Patients will be followed at designated time points along their treatment course to obtain information about ongoing treatment and response, time to tumor progression and overall survival. These parameters will be used in correlational analysis with the metabolic phenotype.

DETAILED DESCRIPTION:
The study is designed to obtain tumor samples from patients undergoing clinically indicated surgical resection of a brain tumor or primary non-CNS tumor after infusion of 13C-glucose, 13C-acetate or 13C-glucose and 13C-acetate. Patients with a brain mass identified on brain imaging and who need surgical resection of the mass will be eligible for this metabolism study. Eligible study patients will be screened, recruited, and enrolled at UT Southwestern Medical Center in the Harold C. Simmons Comprehensive Cancer Center, University Hospital - Zale Lipshy and University Hospital - St. Paul, Children's Medical Center of Dallas as well as at Parkland Health and Hospital System. We will consent 60 patients, including projected screen failures and early withdrawals, and anticipate that we will study 25 patients in this clinical protocol. Once enrolled, patients will undergo a series of preoperative brain imaging studies including 3T MRI with Diffusion Tensor Imaging (DTI) and 1H-MR spectroscopy, 7T MRI and a brain 18FDG-PET scan within 7-14 days of the scheduled operation. Of these studies, only the 3T MRI is standard of care. The DTI and 1H-MR spectroscopy are additional scanning sequences that are being done for research purposes. Similarly, the 7T MRI and the 18FDG-PET are being done for research purposes only. On the day of surgery, the patient will have a peripheral IV started while waiting in the preoperative holding area and a 20% solution of either [U-13C]glucose and/or [1,2-13C]acetate (to be determined for each individual patient by the PI) will be infused at a rate of 4g/hr for a maximum of 4 hours. During the infusion period, 4 timed blood samples will be collected for NMR analysis of 13C-glucose in the blood. The infusion will continue until the tumor has been resected and samples have been collected and flash frozen for 13C-NMR spectral analysis and molecular analyses. The infusion and tumor collection for 13C-NMR analysis is being done for research purposes only. However, the remainder of the neurosurgical operative and post-operative procedures will be followed according to standard practice. The patient will be seen 10-14 days after surgery for a follow up visit at which time an assessment of adverse events will be performed. Thereafter, every 6 months for 5 years or until death, the patient will be contacted and data regarding treatment, responses, and tumor progression will be collected for correlative analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, any age and any racial or ethnic group
* Spanish-speaking patients will be eligible
* Pre-operative brain MR imaging suggestive of a brain tumor or pre-operative imaging showing a tumor or biopsy of a tumor mass prior to planned resection of the mass
* Patient able and willing to provide informed consent or Legal parent or guardian willing and able to provide informed consent for patient under age 18.
* Karnofsky Performance status > 70%
* Negative serum pregnancy test or child bearing potential terminated by surgery, radiation, menopause or current use of two approved methods of birth control

Exclusion Criteria:

* Patient or legal parent/guardian unable to provide informed consent
* Karnofsky Performance status < 70%
* Patients who are claustrophobic or have other contraindications to MRI, such as impanted pacemaker device vascular clips, surgical clips, prosthetic valves, pacemakers, otologic implants
* NYHA class III and IV congestive heart failure
* Psychiatric or addictive disorders that preclude obtaining informed consent
* Unstable angina
* Pregnant or lactating women
* Women of childbearing potential who refuse a pregnancy test (performed during screening)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-08 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
metabolic phenotype correlation to clinical endpoints | at end of follow-up period- between days 1-14
  To correlate the metabolic phenotype obtained from histopathological diagnosis with the clinical endpoints of time to tumor progression and overall survival during the 5 years of patient follow-up

SECONDARY OUTCOMES:
baseline imaging data review | at time of study entry- within 14 days of surgery
  To compare and contrast baseline imaging data obtained on the 7T MR among the major brain tumor histological subtypes (e.g. low grade gliomas, glioblastoma, brain metastases) with emphasis on the differences in vascular integrity and extent of tumor infiltration for each subtype
molecular profiling | after surgical resection- day 0
  To correlate changes on 7T with the molecular profile of the primary resected tumor (molecular profiling is being done under a separate IRB approved protocol).

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Maher, MD, PhD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Southwestern, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No